CLINICAL TRIAL: NCT01317186
Title: The Role of FGF23 and Asymmetric Dimethylarginine (ADMA) in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Bülent Huddam, Ankara Education and Research Hospital
Other Study IDs: NEPH002
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Metabolic Diseases; Chronic Kidney Disease
Keywords: FGF 23; ADMA; chronic kidney disease; Ca-P metabolism disorder
MeSH Terms: conditions — Metabolic Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group I: Stage 2 Non-diabetic Chronic Kidney Disease
- Group II: Stage 3 Non-diabetic Chronic Kidney Disease
- Group III: Stage 4 Non-diabetic Chronic Kidney Disease

SUMMARY:
In chronic kidney disease calcium (Ca) and phosphate (P) metabolism disorders are very common and also they are one of the leading causes of morbidity in these population. FGF23 is a novel factor that contributes Ca-P disorders. It has been hypothesized that FGF 23 increase is mediated by asymmetric dimethylarginine (ADMA). The aim of the study is to evaluate this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* between ages of 18 - 65 years old
* chronic kidney disease of stage 2-4

Exclusion Criteria:

* presence of diabetes mellitus or ischemic hearth disease
* taking vitamin d therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 2-4 Non-diabetic Chronic Kidney Disease patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Education and Research Hospital, Ankara, Turkey (Türkiye)